CLINICAL TRIAL: NCT00021970
Title: Modifying Oxidative Damage in WAVE - Ancillary to WAVE
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 979; R01HL068397 (NIH)
Record Dates: First submitted 2001-08-10; First posted 2001-08-10 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
To determine the effects of four treatments (placebo, a vitamin E and C regimen, a hormone replacement regimen, and a combined vitamin/hormone replacement regimen) on specific markers of oxidative damage in coronary arteries of postmenopausal women.

DETAILED DESCRIPTION:
BACKGROUND:

Supplemental vitamin E has been associated with a reduced risk of recurrent myocardial infarctions, with efficacy related to dosage and the duration of treatment. Its effects may be enhanced by vitamin C, an antioxidant that can regenerate vitamin E activity. Theoretically vitamin E and C (VitE/C) accumulate in the vascular wall with a concurrent reduction in oxidative damage, a primary feature of atherosclerotic lesions. Estrogen/hormone replacement therapy (HRT) also may reduce oxidative damage, and it may enhance the effect of vitamin E and C. These hypotheses are supported by studies defining oxidation-dependent accumulation of lipids in developing atherosclerosis; the detection of oxidative damage products, such as oxidized-LDL particles, in human atherosclerotic lesions; and clinical studies associating antioxidant or estrogen supplementation with reductions in oxidative damage cardiovascular disease. Nevertheless, no human studies have evaluated the effect of long-term VitE/C treatment, which has been reported as being the most effective prevention factor by epidemiologic studies, on specific. biochemical markers of oxidative damage and concurrently their association with recurrent cardiovascular disease. In addition, no studies have characterized the effect of long-term HRT on markers of oxidative damage or HRT's potential synergistic effect with VitE/C therapy.

DESIGN NARRATIVE:

The study assayed specific biochemical measures of oxidative damage (all markers at closeout and nitrotyrosine and chlorotyrosine also at baseline) in the Women's Angiographic Vitamin and Estrogen (WAVE) Trial, which randomized 420 38-86 year old women with a prior cardiovascular disease event to placebo, Vitamin E/C, hormone replacement therapy (HRT) or the combination of VitE/C and HRT. WAVE determined the efficacy of these treatments on quantitative angiographic evaluation of minimal coronary artery diameter performed at baseline and at the final visit to be completed during the first 10 months of 2001. The ancillary study measured oxidation products from several classes of compounds (lipids by F2-isoprostanes, proteins by nitrotyrosine and chlorotyrosine, and DNA by 8-hydroxy-2'-deoxyguanosine), thereby studying several major pathways that may lead to atherogenesis. In addition, inflammation with C-reactive protein, platelet activation with p-selectin, altered lipid metabolism with a lipid profile and other characteristics of the study population were integrated into the assessment of oxidative damage in WAVE. By measuring these various factors and by assessing oxidative damage in several classes of compounds, the authors tested the relationships among specific pathways of oxidative damage, supplemental VitE/C and/or HRT and other risk factors upon the progression of established macrovascular disease.

ELIGIBILITY:
No eligibility criteria

Ages: 38 Years to 86 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-04; Study Completion 2005-03

CONTACTS AND LOCATIONS:
Overall Officials: Michael Steffes — University of Minnesota